CLINICAL TRIAL: NCT05328479
Title: The Study of Treatment Outcome and Immunogenicity of mild-to Moderate COVID-19 Patients During the Delta vs. the Omicron Pandemic
Brief Title: Plasma Immunity of Mild SARS-CoV-2 Omicron and Delta Pandemic in Thailand
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 769/2564(IRB1)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; antibody; immunity; home isolation; vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators assessed the effect of treatment for COVID and immunity of the volunteers who admitted to the home isolation.

DETAILED DESCRIPTION:
The investigators aimed to assess the effect of treatment for COVID and immunity of the volunteers who admitted to the home isolation. The investigators compared the population between the age groups 12-18 years, 18-45 years and over 45 years to monitor the symptoms of coronavirus patients treated in home isolation and long-term symptoms including factors related to the patient's recovery in the past, present, and future.

ELIGIBILITY:
Inclusion Criteria:

1. patient with infected with the novel coronavirus disease 2019 (COVID-19) who has been end of self-quarantine at Siriraj Hospital more than 21 days.
2. Thai nationality, able to read and write Thai language
3. able to use telephone and line to communicate

Exclusion Criteria:

1. people who received additional vaccination after leaving quarantine before the day of the immunization test

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The COVID-19 patients who confirmed by RT-PCR at Siriraj hospital since July 8, 2021 with mild to moderate symptoms and isolated in patients' own home so-called "Siriraj Home isolation".
Sampling Method: Probability Sample
Enrollment: 5181 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 RBD IgG | Baseline
  Anti-RBD IgG (BAU/mL)
Anti-SARS-CoV-2 NP | Baseline
  Anti-SARS-CoV-2 NP (PRNT50 titer)
Cycle threshold of the first PCR test | Baseline
  Cycle threshold (Ct)

SECONDARY OUTCOMES:
Number of vaccine injection | Baseline
  Number of vaccine injection
Type of vaccine injection | Baseline
  Type of vaccine injection

CONTACTS AND LOCATIONS:
Overall Officials: Korapat Mayurasakorn, MD., Principal Investigator — Doctor in Family Medicine
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand